CLINICAL TRIAL: NCT05006625
Title: Implementation of a Collaborative Care Model to Screen and Treat Depression Among Adolescents and Young Adults Ages 15-24 Years Seeking HIV Treatment and Prevention Services in Bangkok, Thailand
Brief Title: Implementation of a Collaborative Care Model to Manage Depression Among Adolescents and Young Adults in HIV Services in Thailand
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Principal Investigator, Wipaporn Natalie Songtaweesin, MD., Principal Investigator, Chulalongkorn University
Other Study IDs: CHIMERA
Record Dates: First submitted 2021-04-20; First posted 2021-08-16 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Depression; HIV
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescents and Young Adults: Adolescents and Young Adults Seeking HIV Treatment and Prevention
  Interventions: Other: Collaborative Care Model
- Service Providers: Service Providers for Adolescents and Young Adults Seeking HIV Treatment and Prevention
  Interventions: Other: Collaborative Care Model

INTERVENTIONS:
Other: Collaborative Care Model — Use of the collaborative care model to screen and deliver care for depression in adolescents and young adults aged 15-24 years seeking HIV prevention and treatment services

SUMMARY:
This study aims to investigate the acceptability and feasibility of the implementation of a collaborative care model (CCM) to screen and treat depression. This model will includes cognitive behavioral therapy (CBT) and useof a task-shifting model to address depression among adolescents and young adults (AYA) who are seeking HIV treatment and prevention services at a hospital in Bangkok, Thailand. Analyses will be guided by the consolidated framework for implementation research (CFIR), which will include the identification of facilitators and barriers to implementation of this CCM.

In the last 3 years, 10-20% of AYA patients at King Chulalongkorn Memorial Hospital (KCMH) who seek HIV treatment or prevention services suffer from mental health disorders. As a result, CCM integration for depression screening and treatment was implemented at the 'CU Buddy Clinic' KCMH with the ultimate goal of increasing access to and engagement in mental healthcare with a goal to improve the overall quality of life for Thai AYA. This project will inform a future implementation science study that will focus on how the optimization of integrated mental healthcare into routine AYA HIV treatment and prevention services can impact health outcomes for patients, including ART adherence and long-term viral suppression (AYA living with HIV) and HIV acquisition risk behaviors and PrEP adherence (AYA at risk for HIV).

ELIGIBILITY:
AYA patients at the CU Buddy Clinic (for both quantitative and qualitative study)

Inclusion criteria

* Aged 15-24 years of age
* Starting or currently receiving HIV treatment and prevention services, which includes any individual or combination receipt of the following services: ART, PrEP, HIV testing, receipt of condoms, HIV risk counselling
* Thai Nationality

Exclusion criteria

• Individuals with a history of, or are currently receiving, mental healthcare at the CU psychiatric clinic or elsewhere

Service providers at CU Buddy Clinic

Inclusion criteria

• Current staff providing care at the CU Buddy Clinic with any active patient interface, such as physicians, nurses, peer navigators, psychologists and psychiatrists

Exclusion criteria

* Staff with less than 3 months duration of service at the CU Buddy Clinic
* Staff who are not affiliated with the CU Buddy Clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Service users aged 15-24 starting or currently receiving HIV treatment and prevention services, which includes any individual or combination receipt of the following services: ART, PrEP, HIV testing, receipt of condoms, HIV risk counselling
  2. Staff providing care at the adolescent HIV treatment and prevention services, with any active patient interface, such as physicians, nurses, peer navigators, psychologists and psychiatrists
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the collaborative care model integration to routine HIV care services | 1 year
  Qualitative assessment - in-depth interviews using semi-structured interview guides individually asking service providers and adolescent service users the feasibility of using the collaborative care model on integration of screening and treatment for depression (including CBT) for standard AYA HIV treatment and prevention services, audio recorded, transcripted and coded for qualitative analysis
Acceptability of using the collaborative care model integration to routine HIV care services | 1 year
  Qualitative assessment - in-depth interviews using semi-structured interview guides individually asking service providers and adolescent service users the acceptability of using the collaborative care model on integration of screening and treatment for depression (including CBT) for standard AYA HIV treatment and prevention services, audio recorded, transcripted and coded for qualitative analysis
Facilitators of using the collaborative care model integration to routine HIV care services | 1 year
  Qualitative assessment - in-depth interviews using semi-structured interview guides individually asking service providers and adolescent service users the facilitators of using the collaborative care model on integration of screening and treatment for depression (including CBT) for standard AYA HIV treatment and prevention services, audio recorded, transcripted and coded for qualitative analysis
Barriers of using the collaborative care model integration to routine HIV care services | 1 year
  Qualitative assessment - in-depth interviews using semi-structured interview guides individually asking service providers and adolescent service users the barriers of using the collaborative care model on integration of screening and treatment for depression (including CBT) for standard AYA HIV treatment and prevention services, audio recorded, transcripted and coded for qualitative analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No